CLINICAL TRIAL: NCT01818219
Title: Effects of Abnormal Respiratory Mechanics and Assisted Mechanical Ventilation on Neuro Regulation of Respiration
Brief Title: Effects of Abnormal Respiratory Mechanics and Assisted Mechanical Ventilation on Neuro-regulation of Respiration
Acronym: RegAIN
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Only half recruitment : restrictive respiratory mechanics group not achievable for technical problems
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2012/12; 2012-A01473-40 (Other: IDRCB number (ANSM))
Record Dates: First submitted 2013-02-28; First posted 2013-03-26 (Estimated); Last update posted 2014-11-25 (Estimated); Status verified 2014-11

CONDITIONS: Neuroregulation of Breathing
Keywords: Electrical activity of the diaphragm; Neuro regulation of breathing; Abnormal respiratory mechanics; Assisted mechanical ventilation; Pressure support; Neurally adjusted ventilatory assist

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Study (Experimental)
  Interventions: Procedure: Records of EADI derived parameters

INTERVENTIONS:
Procedure: Records of EADI derived parameters

SUMMARY:
Due to recent technological improvements, it is now possible to record the electrical activity of the diaphragm (Eadi), a direct expression of the central nervous system respiratory center activity. By providing a relatively easy-to-use technique to record Eadi the NAVA (Neurally Adjusted Ventilatory Assist) technology offers a new opportunity to explore the effects of various interventions on neural inspiratory activity in human subjects during spontaneous and assisted ventilation both for normal and simulated abnormal respiratory mechanics.

The main aim of this project is to measure and compare the components of Eadi signal, the direct reflect of the respiratory centers activity, under various conditions of normal and simulated altered respiratory mechanics (either obstructive or restrictive respiratory mechanics° in order to better understand the neuroregulation of breathing. The second aim of the present project is to perform a similar analysis regarding the effects of various modes (Pressure Support and NAVA) and various levels of assisted ventilation both in case of normal and abnormal respiratory mechanics. Based on the information recorded on Eadi and flow and pressure signals, the last aim of this project is to correlate Eadi and pneumatic derived parameters both during spontaneous breathing and assisted ventilation.

Practically, by using the NAVA recording technology, the investigators will perform a physiological study on normal volunteers to explore the effects of normal and simulated abnormal respiratory mechanics on Eadi, flow and pressure signals (airway, oesophageal and transdiaphragmatic pressures) in order to better understand the neuroregulation of breathing. Thirty healthy volunteers with documented normal lung function tests will be included in the study (obstructive respiratory mechanics will be simulated in 15 healthy volunteers and respiratory mechanics will be simulated in 15 healthy volunteers).

ELIGIBILITY:
Inclusion Criteria:

* Man ;
* Less than 35 years old ;
* Non obese (BMI <30 kg/m2) ;
* Normal pulmonary function tests (vital capacity and forced expiratory volume in one second in the normal range for the age and size)
* No history of respiratory disease (asthma, pneumothorax) ;
* No contraindication for nasogastric tube placement

Exclusion Criteria:

* Active or past respiratory disease ;
* Contraindication to nasogastric tube placement ;
* Less than 18 years old;
* Subject protected by the law (eg subject incapable of discernment, wardship subject, ...) ;
* Subject not covered by a social security system ;
* Subject with a subordination relationship with a member of the research team.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2013-02; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Eadi-time curve | Continuous recording during about 6 hours
  Eadi time curve will be recorded. From this curve, several values will be determined for each respiratory cycle: Maximal Eadi value, area under the curve of Eadi, neural inspiratory time and Eadi slope will be measured

SECONDARY OUTCOMES:
Gastric pressure-time curve | Continuous recording during about 6 hours
Oesophageal pressure-time curve | Continuous recording during about 6 hours
Pressure-time curve | Continuous recording during about 6 hours
  Pressure-time curve will be recorded. From this curve, several values will be determined for each respiratory cycle: Maximal inspiratory value and mean airway pressure

CONTACTS AND LOCATIONS:
Locations (1):
- Medical Intensive Care Unit, University Hospital of Angers, Angers, France

REFERENCES:
- [Derived] Piquilloud L, Beloncle F, Richard JM, Mancebo J, Mercat A, Brochard L. Information conveyed by electrical diaphragmatic activity during unstressed, stressed and assisted spontaneous breathing: a physiological study. Ann Intensive Care. 2019 Aug 14;9(1):89. doi: 10.1186/s13613-019-0564-1. PMID 31414251